CLINICAL TRIAL: NCT03677583
Title: Tolerance of Regular Intake of Duckweed Based Food Products
Brief Title: Duckweed Intake Study
Acronym: DIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: NL66051.081.18
Record Dates: First submitted 2018-09-06; First posted 2018-09-19 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-09

CONDITIONS: Gastrointestinal Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Duckweed (Experimental): daily lunch with 150-180g wet weight duck weed
  Interventions: Other: Duckweed
- Spinach (Active Comparator): daily lunch with 150-180g wet weight spinach
  Interventions: Other: Spinach

INTERVENTIONS:
Other: Duckweed — various meal products such as meal soup, quiche, mashed potato, curry and pasta sauce
  Arms: Duckweed
Other: Spinach — various meal products such as meal soup, quiche, mashed potato, curry and pasta sauce
  Arms: Spinach

SUMMARY:
The study aims to study the impact of frequent intake of 150-180 gram duckweed on gastrointestinal complaints and several other health related biomarkers. The study has a randomised parallel design. Two different treatments will be evaluated e.g. a 11-day intervention with duckweed based meals and a 11-day intervention with control/spinach meals. At the start and at the end of the intervention we will collect a blood sample and a urine samples. Questionnaires about gut complaints, stool consistency and frequency, wellbeing, health complaints or other adverse effects will be collected daily during intervention and up to two days after the intervention.

DETAILED DESCRIPTION:
The study aims to study the impact of frequent intake of 150-180 gram duckweed on gastrointestinal complaints and several other health related biomarkers.

Objective: The primary objective is to investigate gastro-intestinal complaints during 11 day duckweed consumption. Secondary objectives are to assess blood based parameters related to general health and urine based biomarkers for kidney function and to investigate consumer acceptance.

Study design: The study has a randomised parallel design. Two different treatments will be evaluated e.g. a 11-day intervention with duckweed based meals and a 11-day intervention with control/spinach meals. At the start and at the end of the intervention we will collect a blood sample and a urine samples. Questionnaires about gut complaints, stool consistency and frequency, wellbeing, health complaints or other adverse effects will be collected daily during intervention and up to two days after the intervention.

Study population: We aim to include 24 healthy volunteers aged 18-50 years. Intervention: A 11-day intervention in which subjects will receive a daily lunch with 150-180g wet weight duck weed or spinach. Products will be incorporated in food products such as pasta, curry, soup etc.

Main study parameters/endpoints: The main study parameter is frequency and severity of gastro-intestinal complaints. Secondary outcomes are intestinal health parameters derived from blood and urine samples taken before and after the intervention.

ELIGIBILITY:
Inclusion criteria

* Apparently healthy men and women
* Age between 18 and 50 years
* Body mass index (BMI) between 18.5 and 24.9 kg/m2

Exclusion criteria

* Any metabolic, gastrointestinal, inflammatory or chronic disease (such as diabetes, anaemia, hepatitis, cardiovascular disease)
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Kidney dysfunction (self-reported)
* Use of medication that may influence the study results, such as gastric acid inhibitors or laxatives
* Reported slimming, medically prescribed or vegan/vegetarian diet
* Current smokers
* Alcohol intake ≥4 glasses of alcoholic beverages per day
* Pregnant, lactating or wishing to become pregnant in the period of the study (self-reported)
* Abuse of illicit drugs
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the department Consumer Science & Health group of Wageningen Food & Biobased Research

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
change in gastro-intestinal complaints | Daily, during 11 days of duckweed intake and up to three days after intake. By questionnaires and Visual Analogue Scale (VAS) scores; from no complains (minimal) to serious complains (maximum)). Higher values represent a worse outcome
  bloated feeling, belching, abdominal pain, flatulence, nausea, diarrhoea, constipation measured via Visual Analogue Scale (VAS)

SECONDARY OUTCOMES:
change in blood hemoglobin | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood glucose | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood Fe (Iron) | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood leukocyte cell counts | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood ALAT | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood GGT | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood eGFR | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood creatinine | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood CRP | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in blood zonulin | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  under fasting conditions
change in urinary biomarkers of health | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  oxalic acid
change in blood pressure | before (D=0) and after (D=11) 11 days of duckweed or spinach intake
  systolic and diastolic bloodpressure

OTHER OUTCOMES:
fiber, fruit and vegetable intake | before the intervention (D=0), this questionaire provides insights in energy and macronutrient consumption
  via a food frequency questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Diederik Esser, Dr, Principal Investigator — Wageningen research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No
will not be shared